CLINICAL TRIAL: NCT01055106
Title: A Multicenter, Randomized, Investigator-Blinded, Phase 2, Dose Ranging Study of Metronidazole Vaginal Gel in the Treatment of Bacterial Vaginosis
Brief Title: Dose Ranging Study of Metronidazole Vaginal Gel in the Treatment of Bacterial Vaginosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Graceway Pharmaceuticals, LLC (Industry)
Responsible Party: Sharon F. Levy, MD / Vice President Product Develpoment, Graceway Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GW05-0904
Record Dates: First submitted 2010-01-21; First posted 2010-01-25 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2011-06

CONDITIONS: Vaginosis, Bacterial; Vaginal Infection
Keywords: bacterial vaginosis; vaginal infection; vaginal discharge; vaginal disease
MeSH Terms: conditions — Vaginosis, Bacterial; Vaginitis; Vaginal Discharge; Vaginal Diseases | interventions — Metronidazole

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1D (Active Comparator)
  Interventions: Drug: GW05
- 3D (Active Comparator)
  Interventions: Drug: GW05
- 5D (Active Comparator)
  Interventions: Drug: GW05
- Metronidazole (Active Comparator)
  Interventions: Drug: Metronidazole

INTERVENTIONS:
Drug: GW05 — vaginal gel once daily regimen A
  Arms: 1D
Drug: GW05 — vaginal gel once daily regimen B
  Arms: 3D
Drug: GW05 — vaginal gel once daily regimen C
  Arms: 5D
Drug: Metronidazole — vaginal gel 0.75% once daily for 5 days
  Arms: Metronidazole

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of GW05 administered in 3 regimens versus metronidazole 0.75% for the treatment of bacterial vaginosis.

DETAILED DESCRIPTION:
This is a multicenter, randomized, investigator-blinded, phase 2, dose ranging study of GW05 vaginal gel administered in 3 regimens compared to metronidazole 0.75% (QD x 5 days) for the treatment of bacterial vaginosis. Subjects will be evaluated at three timepoints (1 screening/baseline visit, post-treatment phone call and 1 test-of-cure visit). The total study duration may be up to 30 days for a subject.

Study medication will be applied intravaginally once daily at bedtime according to the assigned dosing schedule using the supplied 5-gram vaginal applicators.

Investigator blinding will be ensured by utilizing an independent drug dispensing coordinator at each site.

Bacterial vaginosis (BV) is an infection of the vagina (birth canal) that is the result of an overgrowth of bacteria that are often normally found in the vagina. This type of vaginal infection typically does not cause irritation. The most common complaint of patients who suffer from BV is a fishy-smelling vaginal discharge. The amount of vaginal discharge may or may not be increased above a normal discharge. The bad odor may get worse after sexual intercourse or during the menstrual period. BV is also strongly associated with problems during pregnancy, such as premature (early) birth, and with an increased risk of sexually transmitted diseases. Therefore, it is important to treat the infection.

ELIGIBILITY:
Inclusion Criteria:

* Females at least 18 years of age
* In good general health
* Confirmed current diagnosis of bacterial vaginosis (determined at study screening)
* Negative pregnancy test (for women who are able to become pregnant)
* Must abstain from sexual intercourse throughout the first 7 days of thes study
* Must abstain from alcohol ingestion during the treatment period and for one day afterward
* Must not use intra-vaginal products for the duration of the study

Exclusion Criteria:

* Pregnant, lactating, or planning to become pregnant during the study period
* Menstruating at the time of the diagnosis or anticipate the onset of menses during the treatment phase of the study
* Had a medical event within 90 days of the visit (e.g., stroke, heart attack, etc.)
* Received specific treatments/medications /therapy within the designated time period prior to study enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
proportion of subjects with therapeutic cure | day 21 to day 30

CONTACTS AND LOCATIONS:
Overall Officials: Sharon F Levy, MD, Study Director — Graceway Pharmaceuticals
Locations (20):
- United States (20):
  - Women's Health Research, Phoenix, Arizona
  - Precision Trials, Phoenix, Arizona
  - NEA Women's Clinic, Jonesboro, Arkansas
  - Women's Health Center Inc, San Diego, California
  - Downtown Women's Healthcare, Denver, Colorado
  - Miami Research Associates, Miami, Florida
  - Segal Institiute for Clinical Research, North Miami, Florida
  - All Women's Healthcare of West Broward, Plantation, Florida
  - Atlanta North Gynecology, Roswell, Georgia
  - Women's Health Practice, Champaign, Illinois
  - ActivMed Practices & Research, Haverhill, Massachusetts
  - Grand Rapids Women's Health, Grand Rapids, Michigan
  - Saginaw Valley Medical Research Group, Saginaw, Michigan
  - Women's Health Research Center, Plainsboro, New Jersey
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Jackson Clinic, Jackson, Tennessee
  - Adams Patterson OBGYN, Memphis, Tennessee
  - Women's Partners in Health, Austin, Texas
  - TMC Life Research, Houston, Texas
  - Tidewater Physicians for Women, Norfolk, Virginia

REFERENCES:
- [Derived] Chavoustie SE, Jacobs M, Reisman HA, Waldbaum AS, Levy SF, Hillier SL, Nyirjesy P. Metronidazole vaginal gel 1.3% in the treatment of bacterial vaginosis: a dose-ranging study. J Low Genit Tract Dis. 2015 Apr;19(2):129-34. doi: 10.1097/LGT.0000000000000062. PMID 24983350